CLINICAL TRIAL: NCT03839355
Title: Randomized Trial of Apixaban vs Dose Adjusted Warfarin in Reducing Rate of Cognitive Function Decline, Silent Cerebral Infarcts and Cerebral Microbleeds in Non-valvular Atrial Fibrillation Patients With CHA2DS2-VaSc Score = 2
Brief Title: Trial of Apixaban vs Warfarin in Reducing Rate of Cognitive Decline, Silent Cerebral Infarcts and Cerebral Microbleeds in Patients With Atrial Fibrillation
Acronym: ARISTA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to slower than anticipated enrollment.
Sponsor: Mayo Clinic (Other)
Collaborators: Pfizer (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Malini Madhavan, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 17-010544
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Atrial Fibrillation
Keywords: Apixaban; Warfarin
MeSH Terms: conditions — Atrial Fibrillation | interventions — apixaban; Warfarin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eliquis (Active Comparator)
  Interventions: Drug: Apixaban
- Warfarin (Active Comparator)
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Apixaban — Dosage either 5mg or 2.5mg for 2 years
  Other Names: Eliquis
  Arms: Eliquis
Drug: Warfarin — Dosage assessed by your treating physician for 2 years
  Other Names: Coumadin
  Arms: Warfarin

SUMMARY:
The investigators' central hypothesis is that in patients with atrial fibrillation, anticoagulation with Apixaban reduces the rate of decline in cognitive function, when compared to Warfarin. The investigators also hypothesize that Apixaban reduces cognitive decline by reducing the rate of new cerebral infarction and cerebral microbleeds detected by cerebral MRI compared to warfarin.

ELIGIBILITY:
Inclusion Criteria:

* Non-valvular Atrial Fibrillation
* CHA2DS2-VASc Score > or = to 2
* Never been treated with Apixaban (Eliquis) or prior treatment of < 1 month
* Candidate for oral anticoagulation as assessed by a treating physician

Exclusion Criteria:

* Valvular Atrial Fibrillation (Rheumatic valve disease,Moderate or greater mitral stenosis,Mechanical cardiac valve)
* Active Bleeding
* Prior treatment with Apixaban >1 month
* Recent stroke within 7 days
* Dementia
* Implanted devices not compatible with MRI/any cardiac implanted device
* Claustrophobia
* Active alcohol/drug abuse
* Life expectancy < 1 year
* Taking asprin with >100mg doses
* Known hypersensitivity to warfarin or Apixaban
* Severe renal insufficiency
* Prior severe bleeding (Intracranial bleeding (subdural, subarachnoid, intraparenchymal bleeding),GI bleed requiring transfusion,Bleeding from other sites requiring transfusion)
* Psychosocial reasons that make study participation impractical
* Currently enrolled in another IND or IDE trial that has not completed the primary endpoint or that clinically interferes with the current study endpoints
* Co-morbid condition(s) that could limit the subject's ability to participate in the trial or to comply with follow-up requirements, or that could impact the scientific integrity of the study.
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either psychiatric or physical illness
* Current or expected systemic treatment with strong dual inhibitors of CYP3A4 and P-gp (Any one of rifampin, carbamazepine, phenytoin, St. John's Wort, ketoconazole, itraconazole, ritonavir, clarithromycin)
* Need for dual anti-platelet therapy with aspirin and another agent such as thienopyridine

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malini Madhavan, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eliquis | Warfarin
Started | 18 | 16
Completed | 17 | 16
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eliquis | Warfarin | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.4 (5.84) | 76.4 (5.61) | 76.9 (5.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 11 | 7 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: Standardized Neurocognitive Function Score
Description: Assess the change in cognitive function using standardized neurocognitive assessment.
Time Frame: Baseline, Year 1, Year 2
Population: Study terminated due to slower than anticipated enrollment. Data was not collected or analyzed.
Arm/Group | Eliquis | Warfarin
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: MRI Evidence of Silent Cerebral Infarct
Description: Magnetic Resonance Imagining of the brain to assess the development of new silent cerebral infarcts.
Time Frame: Baseline, Year 2
Population: Study terminated due to slower than anticipated enrollment. Data was not collected or analyzed.
Arm/Group | Eliquis | Warfarin
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: MRI Evidence of New Cerebral Micro-bleeds
Description: Magnetic Resonance Imagining of the brain to assess the development of new cerebral micro-bleeds
Time Frame: Baseline, Year 2
Population: Study terminated due to slower than anticipated enrollment. Data was not collected or analyzed.
Arm/Group | Eliquis | Warfarin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of treatment for approximately 24 months.
Arm/Group | Eliquis | Warfarin
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 0/18 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT03839355/Prot_SAP_000.pdf